CLINICAL TRIAL: NCT01325467
Title: Detection of Coronary Artery Disease Using Analysis of High Frequency QRS: The HyperQ Registry
Acronym: HyperQ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BSP Biological Signal Processing Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Clin_05_01
Record Dates: First submitted 2011-03-28; First posted 2011-03-29 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; high frequency QRS analysis; ischemia; exercise testing; diagnosis of coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease; Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This will be a registry study that will enroll patients referred for an ECG treadmill test with nuclear myocardial perfusion imaging (MPI). The high frequency QRS (HFQRS) information will be recorded and analyzed automatically and simultaneous with the standard ECG signals by the HyperQ System. Results of subsequent tests performed on each patient will be collected and used to enhance the reliability of designating each patient as a CAD-negative (i.e., no significant coronary artery disease) or a CAD-positive (i.e., significant coronary artery disease).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Referred for exercise MPI due to suspected coronary artery disease

Exclusion Criteria:

* Acute Coronary Syndrome (Unstable angina/NSTEMI/STEMI)
* Pre-excitation syndrome
* QRS duration > 120 ms
* Atrial Fibrillation or significant ventricular arrhythmia
* Treatment with Digoxin
* Pacemaker with 100% pacemaker dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients referred for an exercise ECG treadmill test with nuclear myocardial perfusion imaging (MPI).
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
CAD status | one month follow up
  The main goal of this registry will be to compare sensitivity, specificity, positive and negative predictive values of the HyperQ HFQRS analysis for detecting the presence of coronary artery disease to that of standard ECG analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jamieson M Bourque, MD, Principal Investigator — University of Virginia Health System; Robert Schwartz, MD, Principal Investigator — Minneapolis Heart Institute Foundation
Locations (3):
- United States (3):
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Virginia, Charlottesville, Virginia